CLINICAL TRIAL: NCT01860235
Title: Topical Intrapocket Anesthesia With Prilocaine and Lidocaine as Alternative to Injectable Anesthesia During Scaling and Root Planing - A Randomized Clinical Trial
Brief Title: EMLA Topical Anesthetic During Scaling and Root Planing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franciscan University Center (Other)
Responsible Party: Principal Investigator, Raquel Pippi Antoniazzi, Topical intrapocket anesthesia with prilocaine and lidocaine as an alternative to injectable anesthesia during scaling and root planing - A randomized clinical trial, Franciscan University Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EMLA2012
Record Dates: First submitted 2013-05-08; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Local Anesthesia; Pain, Postoperative; Self-Perception
Keywords: Local anesthesia; Pain measurement; Pain perception; Dental anesthesia; Root planing
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine, Prilocaine Drug Combination; Benzocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- sextant 1 (Experimental): Treatment with subgingival scaling and root planing was done in 6 weekly sessions, being the sextant 1 in the randomization for experimental procedures (EMLA)
  Interventions: Drug: EMLA
- sextant 2 (Active Comparator): Treatment with subgingival scaling and root planing was done in 6 weekly sessions, being the sextant 1 in the randomization for experimental procedures (Injectable anesthesia)
  Interventions: Drug: Injectable anesthesia
- sextant 3 (Active Comparator): Treatment with subgingival scaling and root planing was done in 6 weekly sessions, being the sextant 1 in the randomization for experimental procedures (2% Benzocaine)
  Interventions: Drug: 2% Benzocaine
- sextant 4 (Placebo Comparator): Treatment with subgingival scaling and root planing was done in 6 weekly sessions, being the sextant 1 in the randomization for experimental procedures (Placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EMLA — % eutectic mixture of 25mg/g lidocaine and 25 mg/g of prilocaine
  Other Names: EMLA®, AstraZeneca, Cotia, SP, Brazil
  Arms: sextant 1
Drug: Injectable anesthesia — Injectable anesthesia 2% lidocaine with epinephrine 1:100.000
  Other Names: Alphacaine®, DFL, Rio de Janeiro, Brazil
  Arms: sextant 2
Drug: 2% Benzocaine — Topical anesthetic - 200mg/g of 2% benzocaine
  Other Names: Benzotop ®, DFL, Rio de Janeiro, Brazil
  Arms: sextant 3
Drug: Placebo — Manipulated with the same appearance and viscosity of topical anesthetics mentioned above
  Other Names: manipulated topical anesthetics
  Arms: sextant 4

SUMMARY:
Injectable anesthesics previous to subgingival scaling and root planing (SRP) presents some disadvantages like fear of the needle insertion, long-lasting effect and prolonged dampening of adjacent tissues. This study will compare the intrapocket anesthetic effectiveness of a skin topical anesthesic EMLA with intrapocket 2% benzocaine, intrapocket placebo and injectable anaesthesia for SRP in a Split-mouth, double-blind, clinical trial study.

DETAILED DESCRIPTION:
Objective: The aim of this study was to compare the effect of a eutectic mixture containing 25 mg/g of lidocaine and 25 mg/g of prilocaine (EMLA®) with injectable 2% lidocaine, topical benzocaine, and 2% placebo for reducing pain during subgingival scaling and root planing (SRP) procedures.

Methods: Thirty-two patients were enrolled in this split-mouth, double-blind randomized clinical trial. Patients were randomized to a sequence of four anesthetics: 25 mg/g lidocaine and 25 mg/g of 5% prilocaine (EMLA®), injectable 2% lidocaine, topical 2% benzocaine, or placebo. Pain and discomfort were measured using a Visual Analogue Scale (VAS) and Verbal Scale (VS). Patient satisfaction with anesthesia was also determined at the end of each treatment session.

ELIGIBILITY:
Inclusion Criteria:

* eligible individuals for the study were selected from those requiring SRP with at least 2 experimental teeth in four of the six sextants.
* each experimental teeth had to present ≥ 1 site with probing depth ≥ 5 mm associated with BP after treatment of gingivitis (without marginal bleeding).
* furthermore, individual should present ≥ 18 years-old, have not ever done periodontal treatment and be able to understand Verbal Scale (VS) and Visual Analog Scale (VAS).

Exclusion criteria:

* patients that related allergy history or sensitivity reaction to any used amide or ester anesthetics form,
* who received anesthesia or sedation 12 hours before SRP,
* who presented ulcerated lesions or abscesses in the oral cavity,
* who presented oral pathologies with immediate surgical,
* who had prior abuse alcohol history, pregnant women,
* who presented uncontrolled hypertension or
* who had participated in a clinical trial of investigational drug before four months from the beginning of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pain and discomfort | For each tooth was evaluated intraoperative pain using the Visual Analog Scale (5 minutes after the start of the instrumentation) and postoperative immediately after instrumentation. At the end of the procedure, was asked Verbal Scale, for 4 weeks.
  For each experimental tooth, the patient was asked to indicate the intensity of pain and discomfort experienced intraoperatively using the VAS (VAStrans) (5 minutes after the start of the instrumentation in each tooth) and postoperatively (VASpost) immediately after the end of instrumentation of the respective tooth. At the end of the procedure, the patient was asked to also describe the pain sensation of the tooth using VS as: no pain (0), mild pain (1), moderate pain (2), severe pain (3), or extremely severe pain (4).

SECONDARY OUTCOMES:
Patient satisfaction with anesthesia | Determined at the end of all treatment sessions, for 4 weeks.
  Patient satisfaction with anesthesia was determined at the end of all treatment sessions using the following four categories: very satisfactory, satisfied, not satisfied, and completely unsatisfactory.
Injectable anesthetic requirement | If pain persisted after this second application, then an anesthesia infiltration/block was performed, for 4 weeks.
  Percentage of subjects injectable anesthesia requirements in different anesthetic groups. In case of occurrence of pain during the subgingival SRP, an additional dose of the same anesthesic was repeated. If pain persisted after this second application, then an anesthesia infiltration/block was performed.
Adverse Events | Determined when each patient returned for the next treatment session, for 4 weeks.
  When each patient returned for the next treatment session, they were asked about the occurrence of pain, discomfort, localized ulceration, edema, or desquamation of the oral mucosa.